CLINICAL TRIAL: NCT06438367
Title: Mass Balance Study of [14C]TGRX-326 in Healthy Adult Chinese Male Participants
Brief Title: TGRX-326 Pharmacokinetic Mass Balance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen TargetRx, Inc. (Industry)
Collaborators: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TGRX-326-1004
Record Dates: First submitted 2024-05-27; First posted 2024-05-31 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: TGRX-326 (Experimental): healthy subjects will be given 60mg/100uCi[14C]TGRX-326 in suspension
  Interventions: Drug: [14C]TGRX-326

INTERVENTIONS:
Drug: [14C]TGRX-326 — Healthy subjects will be given TGRX-326 60 mg orally on day 1.
  Other Names: TGRX-326

SUMMARY:
This is a pharmacokinetic study for TGRX-326 on mass balance to evaluate distribution, metabolism and excretion of TGRX-326, an ALK inhibitor indicated for treatment of Non-small cell lung cancer.

DETAILED DESCRIPTION:
This study is designed as a single-center, single-dose, non-randomized and open-label study. The study will be conducted in healthy male participants to evaluate distribution, metabolic pathways and route of excretion of TGRX-326 using the Carbon-14 labelled isotope of TGRX-326 compound. Safety evaluation will also be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males
* Age between 18 and 45 years old (both limits included)
* Body weight index between 19.0 and 26.0 kg/m2 (both limits included), and body weight not less than 50.0kg
* Willing to consent
* Able to communicate with investigator and complete study according to study protocol

Exclusion Criteria:

* Clinically significant results from comprehensive physical and clinical examinations
* Positive results on hepatitis, HIV or syphilis
* Clinically significant results from eye examination
* Usage of inducer or inhibitor drugs to drug metabolism with 30 days prior to screening
* Usage of any prescription or non-prescription drug, Chinese herbal medicine or dietary supplements
* Presence of any significant medical history or clinical conditions that could affect study results per investigators' judgement
* Presence of any condition that could affect drug absorption
* Reception of major surgery within 6 months before screening, or surgical wounds not completely healed
* Presence of allergic reactions or may be allergic to ingredients in the investigational drug
* Presence of hemorrhoids, or having history of or is having conditions that cause bloody feces
* Habitual congestion or diarrhea
* Alcohol abuse or excessive alcohol consumption within 6 months before screening
* Excessive smoking within 3 months before screening
* Substance abuse or positive results on urine substance test
* Habits of grapefruit juice consumption or excessive caffeinated drinks consumption
* History of long-term exposure under radiation; or significant radiation exposure 1 year before this study; or participation in other radioactive drug studies
* Having difficulties to receive venous needle puncture, or cannot tolerate venous needle puncture, or history of hematophobia or needle sickness
* Participation in any other clinical studies within 3 months before screening
* Reception of vaccine within 1 months before screening, or planning to be vaccinated during the study
* Planning to have children or donate sperms during the study and within 1 year after the study, or Not agreeing to take contraceptive measures during and within 1 year after study completion
* Blood donation or blood loss of > 400 ml within 3 months before screening; blood donation or blood loss of > 200 ml within 1 month before screening; reception of blood transfusion within 1 months before screening, or planning to donate blood within 3 months after study completion
* Having special dietary requirements and unable to follow the uniform dietary plan in the study
* Any conditions that the investigator deemed unfit for the study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2024-06-26 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-07-21 (Actual)

PRIMARY OUTCOMES:
Urine radioactivity | Day-1 (day before dosing), Day 1 to Day 18 after dosing
  [C14]TGRX-326 radioactivity detected in urine
Fecal radioactivity | Day-1 (day before dosing), Day 1 to Day 18 after dosing
  [C14]TGRX-326 radioactivity detected in feces
Plasma AUC (Area under curve) percentage | Day-1 (day before dosing), Day 1 to Day 18 after dosing
  percentage of [C14]TGRX-326 radioactivity in plasma
Urine %Dose | Day-1 (day before dosing), Day 1 to Day 18 after dosing
  percentage of [C14]TGRX-326 radioactivity in urine
Fecal %Dose | Day-1 (day before dosing), Day 1 to Day 18 after dosing
  percentage of [C14]TGRX-326 radioactivity in feces
Plasma Cmax | Day-1 (day before dosing), Day 1 to Day 18 after dosing
  Maximum concentration of [C14]TGRX-326 measured in plasma
Plasma Tmax | Day-1 (day before dosing), Day 1 to Day 18 after dosing
  Time to maximum concentration of [C14]TGRX-326 measured in plasma

SECONDARY OUTCOMES:
Adverse events/serious adverse events | From screening through completion of study, an average of 1 to 1.5 months.
  to record and analyse subjects with adverse events (AEs) and serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Liyan Miao, MD, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No